CLINICAL TRIAL: NCT03351023
Title: Healthful Dietary Patterns and Risk of Hearing Loss in Women
Brief Title: Healthful Diets and Risk of Hearing Loss
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Gary C Curhan, Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2007P000876
Record Dates: First submitted 2017-11-19; First posted 2017-11-22 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nurses' Health Study II: Nurses' Health Study II, an ongoing cohort study of 116,430 female registered nurses in the US, aged 25-42 at enrollment in 1989. Participants have been followed by biennial mailed questionnaires that elicit updated information on diet, lifestyle, and various health outcomes; the follow-up rate over 26 years exceeds 90% of the eligible person-time.
  Interventions: Other: no intervention-this was an observational study

INTERVENTIONS:
Other: no intervention-this was an observational study

SUMMARY:
To prospectively examine the relations between adherence scores for three healthful dietary patterns, the Alternate Mediterranean diet (AMED), the Dietary Approaches to Stop Hypertension (DASH), and the Alternative Healthy Eating Index (AHEI-2010), and risk of hearing loss in the Nurses' Health Study II.

ELIGIBILITY:
Inclusion Criteria:

* The investigators limited the study to women who provided information on their hearing on the 2009 or 2013 questionnaire.

Exclusion Criteria:

* The investigators excluded those who did not provide responses to the hearing questions on either questionnaire, reported a hearing problem that began before baseline for the current analysis (1991) or did not report date of onset, or reported cancer other than non-melanoma skin cancer. The investigators also excluded women who did not complete the baseline diet questionnaire and who had missing diet information for each subsequent time period.

Ages: 27 Years to 66 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: The Conservation of Hearing Study (CHEARS) examines risk factors for hearing loss among participants in the Nurses' Health Study II, an ongoing cohort study of 116,430 female registered nurses in the US, aged 25-42 at enrollment in 1989. Participants have been followed by biennial mailed questionnaires that elicit updated information on diet, lifestyle, and various health outcomes; the follow-up rate over 26 years exceeds 90% of the eligible person-time. After exclusions, a total of 70,966 women were included in the analyses.
Sampling Method: Non-Probability Sample
Enrollment: 70966 (Actual)
Dates: Start 1991-07-01 (Actual); Primary Completion 2013-06-30 (Actual); Study Completion 2013-06-30 (Actual)

PRIMARY OUTCOMES:
Hearing loss | 1991-2013
  The primary outcome, self-reported hearing loss that was moderate or worse in severity, was determined based on responses to the 2009 and 2013 questionnaires on which participants were asked about their hearing. On the 2009 main questionnaire, participants were asked, "Do you have a hearing problem?" (no, mild, moderate, severe), and "At what age did you first notice a change in your hearing?" On the 2013 main questionnaire, participants were asked, "Which best describes your hearing?" (excellent, good, a little hearing trouble, moderate hearing trouble, deaf), and "Have you noticed a change in your hearing?" and, if the response was "Yes," "At what age did you first notice a change in your hearing?"

SECONDARY OUTCOMES:
hearing loss in HSSQ | 1991-2013
  Detailed hearing-related information was collected electronically in 2012 supplemental questionnaire from a representative subcohort of NHS II participants (n= 33,102) with and without reported hearing problems, including information on previous evaluation for hearing loss, laterality (unilateral or bilateral), and identified causes of hearing loss (e.g. ototoxic medications, ear trauma, otosclerosis, cholesteatoma, Meniere's disease, chronic ear infection). Data from the HSSQ were used to conduct sensitivity analyses using more refined case definitions (e.g. excluding known etiologies and unilateral hearing loss).

CONTACTS AND LOCATIONS:
Overall Officials: Gary Curhan, MD, ScD, Principal Investigator — Brigham and Women's Hospital/Harvard Medical School

IPD SHARING:
Plan to Share IPD: No
For investigators who wish to use the investigators' data, the investigators have adopted a data enclave approach to data sharing within the Nurses' Health Study II cohort. Along with a general description of the cohorts and questionnaires that have been used since 1989 (NHS II), guidelines are available upon request for outside users to access the resources of our studies. Typically, an outside user prepares a brief proposal that is reviewed by the Channing investigator group to identify a local investigator to assist the outside investigator. If uncertainty arises as to the merit of a request, the External Advisory Committees makes a final decision. After approval, the investigators facilitate access to our data either through programming support or orientation to the data.